CLINICAL TRIAL: NCT04834219
Title: Effect of Off-Pump and On-Pump Techniques on Oxidative Stress Biomarkers in CABG
Brief Title: Off-Pump and On-Pump Techniques and Oxidative Stress in CABG Surgery
Acronym: CABG
Status: Completed | Type: Observational
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Ökkeş Hakan Miniksar, Assistant Professor, Bozok University
Other Study IDs: 189_2020.01.18_15
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Cerebral Oxygenation; Oxidative Stress; Myocardial Infarction
Keywords: Coronary artery bypass surgery; Oxidative stress; Cerebral oxygenation
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- On-pump CABG: Patients with an on-pump indication by the cardiovascular surgery department will be included in the study.
  Interventions: Procedure: On-Pump CABG; Procedure: Off-Pump CABG
- Off-pump CABG: Patients with an off-pump indication by the cardiovascular surgery department will be included in the study.
  Interventions: Procedure: On-Pump CABG; Procedure: Off-Pump CABG

INTERVENTIONS:
Procedure: On-Pump CABG — Patients who have undergone on-pump Coronary artery bypass grafting (CABG) surgery are planned by the Department of Cardiovascular Surgery.
Procedure: Off-Pump CABG — Patients who have undergone off-pump Coronary artery bypass grafting (CABG) surgery are planned by the Department of Cardiovascular Surgery.

SUMMARY:
CABG (coronary artery bypass graft) surgery is among the most common heart surgeries performed in the heart pump. In CABG surgery, operations performed on the beating heart without the use of CPB (off-pump) are frequently performed (30-60%) (1).

To the best of our knowledge, there has been no study examining cerebral oxygenation values, oxidative stress levels and postoperative results in CABG operations.

DETAILED DESCRIPTION:
CABG (coronary artery bypass graft) surgery is among the most common heart surgeries performed in the heart pump. In CABG surgery, operations performed on the beating heart without the use of CPB (off-pump) are frequently performed (30-60%) (1). Off-pump coronary artery bypass surgery is also called beating-heart surgery, and its purpose is to avoid cardiopulmonary bypass completely without the support of a heart lung machine, thereby avoiding its adverse effects (3-5). It has been reported that the off-pump CPB surgical method is associated with a decrease in the incidence of early stage and major complications compared to the traditional CPB method (2). Exposure to surgical stress leads to autonomic, visceral, and immunological responses, leading to oxidative stress, neurochemical and hormonal abnormalities (3).In addition to the non-physiological hemodynamic conditions that occur during CABG surgery, a significant increase is observed in inflammatory response and oxidative stress biomarkers due to surgical trauma, cardiopulmonary bypass (CPB) and organ reperfusion injury (4).For this reason, it is important to detect the presence and severity of postoperative adverse outcomes after CABG early. To the best of our knowledge, there has been no study examining cerebral oxygenation values, oxidative stress levels and postoperative results in CABG operations.

This prospective observational study is planned to include 64 adult patients aged 30-80 years who will undergo CABG surgery. Patients will be grouped according to the surgical technique (on-pump and off-pump) determined (indicated) according to the cardiovascular risk status of the patient by the Cardiovascular Surgery department.

Patients' perioperative cerebral hemoglobin oxygen saturations will be recorded with the Regional Oximeter (non-invasive cerebral oxygenation measurement device).

In patients undergoing On-Pump bypass, at the beginning of the CABG surgery (basal), during the aortic clamp, 15 minutes after the clamp is lifted, the remaining 3 ml of blood will be centrifuged at 3000 rpm for 5 minutes and the serum part will be separated.

In off-pump bypass surgery patients, 3 ml of blood will be centrifuged at the beginning of the operation, at the beating phase and 15 minutes after the beating process is completed.

Total antioxidant status, Total oxidant status, Superoxide dismutase, Malondialdehyde will be measured in the Enzyme-Linked ImmunoSorbent Assay device from blood samples taken from all patients in the study, and their concentrations will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Undergo CABG surgery with on-pump and off-pump technique,
* Volunteer to participate in the study,
* 30-80 years old

Exclusion Criteria:

* Those with chronic kidney failure
* Those with liver failure
* Under 30 and over 80

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to participate in this prospective observational study of 64 volunteer patients undergoing Coronary artery bypass grafting (CABG) surgery by the Department of Cardiovascular Surgery.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Oxidative stress level | Intraoperative period
  Oxidative stress biomarker levels between on-pump and off-pump coronary artery bypass groups
TAS | Intraoperative period
  Total antioxidant status
TOS | Intraoperative period
  Total oxidant status
SOD | Intraoperative period
  Superoxide dismutase

SECONDARY OUTCOMES:
Cerebral oximetry | Intraoperative period
  Cerebral haemoglobin oxygen saturations (%)

CONTACTS AND LOCATIONS:
Overall Officials: Ökkeş Hakan Miniksar, Asist.Prof, Study Chair — YOZGAT BOZOK UNIVERSITY
Locations (1):
- Bozok University Medical Center, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hussain G, Azam H, Baig MA, Ahmad N. Early outcomes of on-pump versus off-pump coronary artery bypass grafting. Pak J Med Sci. 2016 Jul-Aug;32(4):917-21. doi: 10.12669/pjms.324.9680. PMID 27648039